CLINICAL TRIAL: NCT06996639
Title: Breaking Fasts Ahead of Cardiac Caths: an Open Label Non-Blinded RCT (BACON-RCT)
Brief Title: Breaking Fasts Ahead of Cardiac Caths
Acronym: BACON-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Samip Vasaiwala, Primary Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY007430
Record Dates: First submitted 2025-04-30; First posted 2025-05-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Stable Angina (SA); Unstable Angina (UA); NSTEMI - Non-ST Segment Elevation MI
Keywords: Fasting; NPO; Cardiac Catheterization; ACS; Angina; Unstable Angina; Worsening Angina; Low Risk NSTEMI; NSTEMI; Acute Coronary Syndrome; Urgent Cardiac Catheterization; Patient satisfaction; Periprocedural care; Non-fasting; Safety outcomes; Pre-procedural protocol; Survey-based research
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; Fasting; Angina Pectoris; Acute Coronary Syndrome; Patient Satisfaction | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): Participants in this group will follow standard pre-procedural fasting guidelines: no solid food for at least 6 hours and no clear liquids for at least 2 hours before their cardiac catheterization or "NPO at Midnight."
  Interventions: Behavioral: Fasting
- Non-Fasting (Experimental): Participants in this group will have no dietary restrictions before their cardiac catheterization and may eat and drink as they normally would.
  Interventions: Behavioral: Non-Fasting

INTERVENTIONS:
Behavioral: Non-Fasting — No pre-procedural fasting required; participants may eat and drink as usual.
  Arms: Non-Fasting
Behavioral: Fasting — Standard pre-procedural fasting (≥6 hours for solids, ≥2 hours for clear liquids) or "NPO at Midnight."
  Arms: Fasting

SUMMARY:
The goal of this clinical trial is to find out whether fasting is necessary before urgent inpatient cardiac catheterizations. For patients presenting with urgent heart-related pain or even mild heart attacks, researchers want to know whether eating and drinking before their procedure improves comfort without raising the risk of complications.

The study will answer:

* Does eating and drinking before the procedure improve patient comfort?
* Does it increase the risk of adverse events like vomiting, aspiration (food or liquid entering the lungs), breathing problems, or death, etc?

Participants will be randomly assigned to either:

* A standard fasting group (no food for 6 hours, no clear liquids for 2 hours), or
* A no-fasting group (able to eat and drink as usual).

Patients will complete brief surveys before the procedure to assess comfort and satisfaction. Researchers will also review medical records weekly and 30 days later to monitor for safety outcomes.

DETAILED DESCRIPTION:
While pre-procedural fasting is a longstanding tradition in cardiac catheterization, there is limited evidence supporting its necessity in low-risk patients undergoing urgent procedures for acute coronary syndromes (ACS). Existing studies have lacked adequate recruitment of ACS patients, comprehensive demographic capture, and long-term outcomes.

This randomized clinical trial will enroll adult inpatients undergoing cardiac catheterization for worsening angina and low risk ACS (unstable angina, and non-high risk NSTEMI's) with planned moderate proceduralist-guided sedation. Participants will be randomized 1:1 to either standard fasting (≥6 hours for solids and ≥2 hours for clear liquids) or no fasting requirement.

The primary endpoint is a composite of patient-reported outcomes assessing comfort and satisfaction. Secondary outcomes focus on clinical safety metrics, such as hemodynamic instability, aspiration pneumonia, ICU admission, procedural sedation requirements, and 30-day mortality, etc.

Proceduralists will remain unblinded; however, outcome assessment and statistical analysis will be performed by blinded third-party personnel. This trial aims to provide high-quality data to assess the necessity and impact of fasting in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* All scheduled urgent inpatient non-high risk cardiac catheterizations for worsening angina (cardiac chest pain or anginal equivalent), unstable angina, or non-high risk NSTEMI-NSTEMI's with GRACE score <140 points) utilizing proceduralist guided sedation

Exclusion Criteria:

* High risk NSTEMI's defined as NSTEMI's with a GRACE score >140 points
* Hemodynamic instability (<SBP 90)
* Unstable arrythmias
* Chest pain refractory to nitroglycerin drip
* New ejection fraction less than 25%
* Evidence of severe decompensated heart failure on presentation requiring BiPAP or mechanical intubation
* Inability to consent
* Patients <18 years old
* Pregnant patients
* Need for general anesthesia
* Acute hypoxic respiratory failure requiring >6L Nasal Cannula Supplementation, BiPAP, or invasive ventilation
* Emergent interventions: STEMI/high risk NSTEMI
* Need for mechanical circulatory support-ECMO, Impella or intra-aortic balloon pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pre-procedural patient satisfaction and comfort | Within one hour pre-cardiac catheterization
  Patient satisfaction and comfort will be assessed using a six-item survey evaluating hunger, thirst, nausea, nervousness, anger, and weakness. Each item is rated on a 5-point Likert scale from 1 ("strongly disagree" = least discomfort) to 5 ("strongly agree" = most discomfort). The total score ranges from 6 (best possible comfort) to 30 (worst possible discomfort). Higher scores indicate greater overall discomfort.

SECONDARY OUTCOMES:
Time since last oral intake | At time of procedure
  Time (in minutes) between last oral intake (food or fluid) as self-reported on pre-procedural survey and start of cardiac catheterization.
Hypotension | During procedure and up to 6 hours post-procedure
  Number of individuals with an occurrence of systolic blood pressure <85 mmHg or mean arterial pressure (MAP) <65 mmHg during or within 6 hours after the procedure.
Hyperglycemia | During or within 6 hours post-procedure
  Number of individuals with an occurrence of blood glucose >200 mg/dL during or within 6 hours after the procedure, based on point-of-care or laboratory testing.
Hypoglycemia | Within 6 hours pre and post-procedure
  Number of individuals with an occurrence of blood glucose <70 mg/dL within 6 hours before, during, or after the procedure based on point-of-care or laboratory testing.
New hypoxic respiratory failure | During or with 6 hours post-procedure, not present prior to catheterization.
  Number of individuals with the development of new hypoxia (SpO₂ <85% on room air or requiring supplemental oxygen >4 L/min) during or within 6 hours post-procedure, not present prior to catheterization.
Aspiration pneumonia | Within 72 hours post-procedure, not present prior to catheterization.
  Number of individuals with a new diagnosis of aspiration pneumonia within 72 hours post-procedure, based on new pulmonary infiltrate on imaging plus clinical signs (e.g., cough, fever, hypoxia), not present prior to procedure.
New non-invasive or invasive ventilation | During or within 24 hours post-procedure
  Number of individuals with the initiation of CPAP, BiPAP, or endotracheal intubation during the procedure or within 24 hours post-procedure.
New intensive care unit (ICU) admission | Within 24 hours post-procedure
  Number of individuals with a new admission to an ICU within 24 hours post-procedure that was not planned prior to catheterization.
Need for emergency surgical intervention | During or within 24 hours post-procedure
  Number of individuals with an unplanned surgical procedure initiated during or within 24 hours after catheterization as a result of a procedural complication.
30-day mortality | 30 days post-procedure
  To be gathered by chart review 30 days post-procedure.
Sedation use | During procedure
  Total volume (mg or mcg) of midazolam and fentanyl administered during the procedure, as documented in the procedural record.

CONTACTS AND LOCATIONS:
Overall Officials: Samip Vasaiwala, MD, Principal Investigator — USF Department of Internal Medicine; Division of Cardiovascular Sciences
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) dataset will include information necessary to support the primary and secondary outcome findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available beginning 3 months and ending 5 years after the publication of results.
Access Criteria: De-identified individual participant data (IPD) will be made available only upon request by ICMJE-affiliated journal editors or peer reviewers during the manuscript review and publication process. Data will not be shared with other external researchers or institutions. The dataset will include information necessary to support the primary and secondary outcome findings.
  No open-access sharing is planned. Requests for IPD must be submitted directly to the principal investigator via email. A data sharing agreement will be required to ensure confidentiality and appropriate use. The study principal investigator and research team will review each request to confirm it originates from a journal editor or peer reviewer and that the purpose aligns with manuscript review or publication.
  Once approved, access will be provided via a secure, encrypted file transfer. All data will be de-identified in accordance with HIPAA standards, and no identifiers will be included.

REFERENCES:
- [Background] Mitchell BK, Tomdio A, Pir MS, Mishra SK, Dayanand P, Bonnet G, Alu MC, Gertz ZM. A Randomized Trial of Cardiac Catheterization With Fasting Versus Liberal Oral Intake: The CALORI Trial. J Soc Cardiovasc Angiogr Interv. 2024 Oct 24;3(12):102291. doi: 10.1016/j.jscai.2024.102291. eCollection 2024 Dec. PMID 39807233
- [Background] Woods C, Wood M, Boylan A, Flanagan ME, Powers J. Fasting Versus a Heart-Healthy Diet Before Cardiac Catheterization: A Randomized Controlled Trial. Am J Crit Care. 2024 Jan 1;33(1):29-33. doi: 10.4037/ajcc2024115. PMID 38161168
- [Background] Saad M, Waqas SA, Aamir J, Sohail MU, Ansari I, Mohan A, Kumar V, Alraies MC. Fasting Versus Nonfasting Before Cardiac Catheterization: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Cardiol. 2025 Mar 1;238:40-46. doi: 10.1016/j.amjcard.2024.11.030. Epub 2024 Nov 28. PMID 39613281
- [Background] Granger CB, Goldberg RJ, Dabbous O, Pieper KS, Eagle KA, Cannon CP, Van De Werf F, Avezum A, Goodman SG, Flather MD, Fox KA; Global Registry of Acute Coronary Events Investigators. Predictors of hospital mortality in the global registry of acute coronary events. Arch Intern Med. 2003 Oct 27;163(19):2345-53. doi: 10.1001/archinte.163.19.2345. PMID 14581255
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Mishra A. Strict versus no fasting prior to cardiac catheterization: a prospective evaluation of safety and clinical outcomes. Can we safely have our patients eat with cardiac catheterization - nix or allow: the CHOW NOW study [abstract 11758].SCAI 2020 Virtual Scientific Sessions: Virtual Conference, May 14 to 16, 2020.
- [Background] Ferreira D, Hardy J, Meere W, Butel-Simoes L, McGee M, Whitehead N, Healey P, Ford T, Oldmeadow C, Attia J, Wilsmore B, Collins N, Boyle A. Safety and care of no fasting prior to catheterization laboratory procedures: a non-inferiority randomized control trial protocol (SCOFF trial). Eur Heart J Open. 2023 Oct 17;3(6):oead111. doi: 10.1093/ehjopen/oead111. eCollection 2023 Nov. PMID 38025651
- [Background] Tamborrino PP, Papi L, Michelotti L, Vitale C, Caravelli P, Petronio AS, Terlizzi E, Della Volpe L, Virlan M, Sardanelli A, Morganti R, De Caterina R. Do We Need Fasting Prior to Coronary Angiography? The CORO-NF Randomized Pragmatic Study. Am J Med. 2024 Jul;137(7):666-672. doi: 10.1016/j.amjmed.2024.01.024. Epub 2024 Feb 7. PMID 38336086